CLINICAL TRIAL: NCT04858399
Title: Examination of Orofacial Muscles With Myotonometer in Obstructive Sleep Apnea Syndrome and Investigation of the Risk of Exposure According to Disease Severity
Brief Title: Muscle Tone Change in Obstructive Sleep Apnea
Acronym: OSASMumecPRO
Status: Completed | Type: Observational
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Tülay Çevik Saldıran, PT, Assistant Professor, Bitlis Eren University
Other Study IDs: BEU_2
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Sleep Apnea Syndromes
Keywords: Muscle Tone; Quality of Life; Depression; Respiration
MeSH Terms: conditions — Sleep Apnea Syndromes; Depression; Respiratory Aspiration | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild Severity OSAS: Mild sleep apnea: An Apnea-Hypopnea Index (AHI) of five to 14 events per hour.
  Interventions: Diagnostic Test: Evaluation
- Moderate Severity OSAS: Moderate sleep apnea: An Apnea-Hypopnea Index (AHI) of 15 to 29 events per hour.
  Interventions: Diagnostic Test: Evaluation
- High Severity OSAS: Severe sleep apnea: An Apnea-Hypopnea Index (AHI) of 30 or more events per hour
  Interventions: Diagnostic Test: Evaluation

INTERVENTIONS:
Diagnostic Test: Evaluation — To examine the differences in respiratory functions, orofacial muscle tone changes, anxiety/ depression, and quality of life of the patients according to the severity of Obstructive Sleep Apnea Syndrome.

SUMMARY:
The study aim of the project is to investigate the differences in respiratory functions, orofacial muscle tone changes, anxiety/depression, and quality of life of the patients according to the severity of Obstructive Sleep Apnea Syndrome. At the same time, to examine the reliability of the use of the MyotonPro evaluation method, which takes place rapidly in the literature and clinic, in the orofacial pharyngeal muscle group.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) syndrome is a common but often unrecognized disorder caused by pharyngeal collapse during sleep and characterized by frequent awakenings, disrupted sleep, and consequent excessive daytime sleepiness. Upper airway resistance increase during sleep and upper airway inspiratory muscle activity decrease especially during bursts of rapid eye movements in REM (Rapid Eye-Movements) sleep. In this study, the differences in respiratory functions, orofacial muscle tone changes, anxiety/depression, and quality of life of the patients according to the severity of Obstructive Sleep Apnea Syndrome will be investigated. The project is planned to be carried out with participants who applied to the Bitlis State Hospital Chest Diseases Clinic and were diagnosed with OSA by polysomnography and other diagnostic methods. Based on "the Apnea-Hypopnea Index OSA rating scoring for adult individuals", participants will be divided into three groups: mild, moderate, and severe OSA. Healthy participants will form the fourth group on the control level. The respiratory functions of the participants will be evaluated with spirometry and a standard application procedure will be used. With the MyotonPro device, the tone of the orofacial muscles (m. digastricus venter anterior and m. mylohyoideus, tongue and m. masseter, m. temporalis) will be evaluated and data transferred to the computer will be reported. In the muscle tonus evaluations, standardization in cervical positioning will be provided by a dual digital inclinometer. The Hospital Anxiety and Depression Scale (HAD) will be used to evaluate the anxiety/depression levels of the participants, and the Short Form-36 (SF-36), which is prescribed as the global gold standard, will be used in the assessment of the quality of life. MyotonPro reliability investigation will be done by two separate researchers. The researchers will perform measurements independently, at the baseline, and after 1 week. MyotonPro evaluations will be based on anatomical localization points. During the measurement, both researchers will use the standard positioning protocol at both evaluation times.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Getting a diagnosis of OSAS with polysomnography.
* Agree to participate in the study.

Exclusion Criteria:

* Having respiratory system disease (COPD, asthma, bronchiectasis, lung cancer, etc.).
* Sedative, hypnotic drug intake. Use of medical supplements such as diazepam.
* Hypothyroidism, acromegaly.
* Diagnosis of a psychiatric illness.
* Uncontrolled arrhythmia causing symptoms or hemodynamic impairment.
* Pulmonary edema.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic in Bitlis.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The muscle tone evaluation | Day 1.
  MyotonPro device will be used for muscle tone evaluation.The device provides a controlled preload of 0.18 N for initial compression of the subcutaneous tissue and then release an additional 15-ms impulse of 0.40 N of mechanical force, which induces a damped or decaying natural oscillation of the tissue35. The calculation formula was as follows: S = amax. mprobe/Δl; amax - maximum amplitude of the oscillation in the acceleration signal; mprobe - mass (preload) of the probe of 0.18 N, Δl - amplitude of the displacement signal.

SECONDARY OUTCOMES:
Evaluation of the anxiety and depression. | Day 1.
  The Hospital Anxiety and Depression Scale will be used to evaluate the anxiety/depression levels of the participants. It consists of two subscales, one measuring anxiety, with seven items, and one measuring depression, with seven items, which are scored separately. Each item was answered by the patient on a 4-point (0 - 3) response category so the possible scores ranged from 0 to 21 for anxiety and 0 to 21 for depression. It takes 2 - 5 min to complete.

OTHER OUTCOMES:
Evaluation of Quality of Life | Day 1.
  The Short Form-36 will be used to evaluate the quality of life of patients. This 36-item, self-administered generic health profile questionnaire provides summary scores in two domains, physical health, and mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis State Hospital, Bitlis, Turkey (Türkiye)